CLINICAL TRIAL: NCT04131972
Title: A Pilot Study of REGENERA Implant in Localized Non- Malignant Breast Lesions Treated by Excision or Lumpectomy
Brief Title: REGENERA Implant in Excised Non-Malignant Breast Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tensive SRL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Tens-BBC/001/2017
Record Dates: First submitted 2019-05-14; First posted 2019-10-18 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Benign Breast Disease
Keywords: Lumpectomy; Bio-absorbable
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm 1 (Experimental): Each patient will be planned to perform 7 study visits and at the second visit excision / lumpectomy and REGENERA implant will be performed during the same surgical intervention.
  Interventions: Device: REGENERA

INTERVENTIONS:
Device: REGENERA — REGENERA breast implant

SUMMARY:
The purpose of this First-in-Human pilot study is to evaluate the safety and performance of REGENERA breast implant in a selected cohort of patients with non- malignant breast lesions treated with excision or lumpectomy in whom the tissue removed is replaced by REGENERA.

DETAILED DESCRIPTION:
This is a pre-market, single center, interventional, open label, non-comparative, pilot first-in-human study on adult female patients with localized non-malignant breast lesion. This study will include an enrollment period of 12 months and 6 months study duration per patient.

The primary objective of this study is to demonstrate the safety profile of a new breast implant (REGENERA) in excision or lumpectomy of non-malignant breast lesions.

The secondary objectives of this study are:

* To assess the safety of the implant procedure
* To assess the feasibility of the implant procedure
* To evaluate the performance of REGENERA breast implant:

  * In replacing the removed tissue
  * In potential interference with current diagnostic standard of care imaging procedures
  * On patient's quality of life and satisfaction
  * On investigator's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 20-85 years
2. Patients eligible for excision or lumpectomy, as per current surgical guidelines
3. Volume deficit compatible with an implant volume of 70 cc
4. Adequate hematopoietic functions
5. Good general health and mentally sound
6. Confirmation of non-malignant lesion (B2 and B3) with no discordance between biopsy and radiological imaging
7. Patients able and willing to give written informed consent form

Exclusion Criteria:

1. Pregnant or breastfeeding women or women who have nursed a child three months within enrolment in the study
2. Non-malignant lesions (B2 and B3) with discordance between biopsy and radiological imaging
3. Infection of the surgical site confirmed pre-operatively by clinical examination
4. Acute or chronic severe renal insufficiency (creatinine values < 180 μmol/L)
5. History of severe asthma or allergies (including to anaesthetics or contrast media)
6. Autoimmune disease
7. Subject with actual concomitant malignancies, lobular neoplasm, metastatic breast carcinoma, sarcoma, malignant phyllodes lesions, or Paget's disease
8. Subject who are known to be carriers of BCRA mutation
9. Inability to undergo MRI or allergy to contrast media
10. Systemic infections in active phase
11. Immunocompromised patients (HIV)
12. Subjects who have participated in another study within the past 3 months
13. Patients who received immunosuppressant therapy in the last 3 months
14. Non-collaborative patients (severe physical disabilities or psychiatric disorders, as per specialist opinion).

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Cumulative number of all Serious Adverse Events | at 6 months from implantion of the device
  Cumulative number of Serious Adverse Events collected throughout the study and associated with the REGENERA implant device (Adverse Device Effects)

SECONDARY OUTCOMES:
Measurement of changes in breast appeareance before and after surgery through antropomorphic chest parameters | at 2 weeks before the implantation of the device (Day 0), 1 week from Day 0, 3 months from Day 0, 6 months from Day 0
  Assess breast appearance before and after surgery with photo and chest measurement. In particular, the following measures, in cm, will be evaluated: sternal notch to nipple (SN), nipple to inframammary fold (NF), nipple to sternum (NM), the areola diameter and the ptosis grade.
Measurement of the reduction of reliability of the currently used diagnostic imaging techniques | at 1 week from the implantation of the device (Day 0), 2 weeks from Day 0, 1 month from Day 0, 3 months from Day 0 and 6 months from Day 0
  Assess the potential interference with current, standard- of-care imaging techniques by evaluation of the following factors: (1) for ultrasound, the possible attenuation of the acoustic beam preventing the visualization of the tissue behind the implant; (2) for magnetic resonance imaging, possible creation, caused by the implant, of images mimicking a pre-invasive or invasive lesion.
Patient Quality of Life measured through Breast-Q questionnaire | at 1 month from the implantation of the device (Day 0), 6 months from Day 0 versus 2 weeks before Day 0
  Measure changes in patient's Quality of Life (QoL) and satisfaction through Breast-Q™ questionnaire (pre- and post-operative Breast Conserving Therapy (BCT) module version 2.0) after surgery versus baseline (prior implantation surgery).
  Breast-Q™ questionnaire includes 7 scales measuring (i) breast satisfaction, (ii) psychosocial well-being, (iii) physical breast well-being, (iv) sexual well-being, (v) patient experience satisfaction with the surgeon, (vi) patient experience satisfaction with the medical equip and (vii) patient experience satisfaction with the hospital staff. Each scale is evaluated by defined questions where the patient has to answer by a numeric scale. For example: "1", "non of the time"; "2", "a little of the time"; "3", some of the time; "4", "most of the time"; "5", "all of the time". Once the questions are answered, a conversion table is applied to convert the raw scale summed score into a score from 0 (worst) to 100 (best).
Patient pain measurement through a Visual Analogue Scale | at 2 weeks before the implantation of the device (Day 0), Day 0, 1 week from Day 0, 2 weeks from Day 0, 1 month from Day 0, 3 months from Day 0 and 6 months from Day 0
  Assess pain intensity with a Visual Analogue Scale (VAS) at each study visit. The VAS measure will be made through a cross (X) that the patient has to put along a bar. The left margin of the bar corresponds to "no pain" (0 score) and the right margin to "worst pain" (10 score).
Measure of the Investigator's satisfaction on the implantation procedure, through a Visual Analogue Scale (VAS) and an ad-hoc questionnaire | implantation satisfaction (VAS + ad-hoc questionnaire) at the implantation of the device (Day 0) and REGENERA performance (VAS) at 6 months from Day 0
  Assess investigator's satisfaction on the implantation procedure, through a Visual Analogue Scale (VAS) and an ad-hoc questionnaire (developed by the Sponsor), and on the REGENERA performance, through a VAS scale.
  The VAS measure will be made through a cross (X) that the patient has to put along a bar. The left margin of the bar corresponds to "no pain" (0 score) and the right margin to "worst pain" (10 score).
  The ad-hoc questionnaire has a unique scale made of 5 levels (1 corresponds to "strongly disagree" and 5 corresponds to "strongly agree") to be used for each question. As there are 12 questions, 12 is the minimum score and 60 is the maximum score as a sum of all answers.
Cumulative number of all Adverse Events associated with the surgical procedure | at 6 months from the implantation of the device
  Cumulative number of all Adverse Events associated with the surgical procedure: number of re-operations and / or explants due to seroma, hematoma, infection, wound dehiscence, skin retraction, acute inflammatory reactions, allergic reactions to the device, persistent pain.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Roncella, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariniello MD, Roncella M, Mazzotta D, Gerges I, Colizzi L, Tamplenizza M, Tocchio A, Martello F, Ghilardi M, Cossu MC, Danti S, Ghilli M. Scaffold-based breast conserving surgery in patients with non-malignant breast lesions: long-term follow-up of a first-in-human pilot study on the REGENERA biomimetic breast implant. Breast Cancer. 2026 Jan;33(1):111-122. doi: 10.1007/s12282-025-01780-w. Epub 2025 Sep 27. PMID 41014462
- [Derived] Mariniello MD, Ghilli M, Favati B, Gerges I, Colizzi L, Tamplenizza M, Tocchio A, Martello F, Ghilardi M, Cossu MC, Danti S, Roncella M. Cell-free biomimetic polyurethane-based scaffold for breast reconstruction following non-malignant lesion resection. A first-in-human study. Breast Cancer. 2023 Jul;30(4):559-569. doi: 10.1007/s12282-023-01446-5. Epub 2023 Mar 28. PMID 36977972